# STATISTICAL ANALYSIS PLAN

Study Code

AZ-RU-00004

Edition Number 3.0

inon i vannoei

Date 6-Aug-2024

A Phase III, Multicentre, Randomized, Double-blind, Single-Dose, 2-Arm, 2-Period, Crossover Study to Investigate the Efficacy of PT027 Compared with Placebo on Exercise-Induced **Bronchoconstriction in Adult Patients with Asthma (BREATH)** 

# **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 8 |
|---|---|---|
| 2 | CHANGES TO PROTOCOL PLANNED ANALYSES | 8 |
| 3 | DATA ANALYSIS CONSIDERATIONS | 8 |
| 3.1 | Timing of Analyses | 8 |
| 3.2 | Analysis Populations | |
| 3.3 | General Considerations | |
| 3.3.1 | General Study Level Definitions | |
| 3.3.1.1 | Period specific post-dose pre-exercise baseline | |
| 3.3.1.2 | Period specific pre-dose baseline | |
| 3.3.1.3 | Average pre-dose baseline | |
| 3.3.1.4 | Absolute and percent change from baseline | 10 |
| 3.3.1.5 | Percentage fall from post-dose pre-exercise baseline FEV <sub>1</sub> | |
| 3.3.1.6 | Crossover difference in maximum percentage fall of FEV <sub>1</sub> | 11 |
| 3.3.2 | Visit Window | 11 |
| 3.3.3 | Handling of Unscheduled Visits | 11 |
| 3.3.4 | Multiplicity/Multiple Comparisons | |
| 3.3.5 | Handling of Protocol Deviations in Study Analysis | |
| 3.3.6 | Missing Data | 12 |
| 4 | STATISTICAL ANALYSIS | 13 |
| 4.1 | Study Population | 13 |
| 4.1.1 | Subject Disposition and Completion Status | |
| 4.1.1.1 | Definitions and Derivations | |
| 4.1.1.2 | Presentation | 14 |
| 4.1.2 | Analysis Sets | |
| 4.1.2.1 | Definitions and Derivations | |
| 4.1.2.2 | Presentation | |
| 4.1.3 | Protocol Deviations | |
| 4.1.3.1 | Definitions and Derivations | |
| 4.1.3.2 | Presentation | |
| 4.1.4 | Demographics | |
| 4.1.4.1 | Presentation | |
| 4.1.5 | Baseline Characteristics | |
| 4.1.5.1 | Presentation | |
| 4.1.6 | Disease Characteristics | |
| 4.1.6.1 | Definitions and Derivations | |
| 4.1.6.2 | Presentation | |
| 4.1.7 | Medical History and Concomitant Disease | |
| 4.1.7.1 | Definitions and Derivations | |
| 4.1.7.2 | Presentation. | |
| 4.1.8 | Prior and Concomitant Medications | |
| 4.1.8.1 | Definitions and Derivations | 16 |
| 41 X / | Presentation | / |

| 4.1.9 | Study Drug Compliance | 18 |
|---|---|---|
| 4.2 | Endpoint Analyses | 18 |
| 4.2.1 | Primary Endpoint. | |
| 4.2.1.1 | Definition | 20 |
| 4.2.1.2 | Derivations. | 20 |
| 4.2.1.3 | Handling of Dropouts and Missing Data | 20 |
| 4.2.1.4 | Primary Analysis of Primary Endpoint | |
| 4.2.1.5 | Sensitivity Analyses of the Primary Endpoint | |
| 4.2.2 | Secondary Endpoint: the percentages of subjects with a maximum | |
| | percentage fall in FEV <sub>1</sub> of <10% and <20% | 22 |
| 4.2.2.1 | Definition | |
| 4.2.2.2 | Derivations | |
| 4.2.2.3 | Handling of Dropouts and Missing Data | |
| 4.2.2.4 | Primary Analysis of Secondary Endpoint | |
| 4.2.2.5 | Supplementary Analysis of Secondary Endpoint | |
| 4.2.3 | Secondary Endpoint: the percentage fall in FEV <sub>1</sub> from post-dose, pre- | |
| | exercise at each timepoint within 60 minutes post-exercise | 22 |
| 4.2.3.1 | Derivations | |
| 4.2.3.2 | Handling of Dropouts and Missing Data | |
| 4.2.3.3 | Primary Analysis of Secondary Endpoint | |
| 4.2.4 | Secondary Endpoint: post-exercise FEV <sub>1</sub> area under the curve from 0 to | |
| | minutes | |
| 4.2.4.1 | Definition | |
| 4.2.4.2 | Derivations | |
| 4.2.4.3 | Handling of Dropouts and Missing Data | |
| 4.2.4.4 | Primary Analysis of Secondary Endpoint | |
| 4.2.5 | Secondary Endpoint: time to recovery | |
| 4.2.5.1 | Definition | |
| 4.2.5.2 | Derivations. | |
| 4.2.5.3 | Handling of Dropouts and Missing Data | 24 |
| 4.2.5.4 | Primary Analysis of Secondary Endpoint | |
| 4.2.6 | Other Endpoints | |
| 4.2.7 | Subgroup Analyses | |
| 4.3 | Pharmacodynamic Endpoint(s) | 25 |
| 4.4 | Pharmacokinetics | |
| 4.5 | Immunogenicity | 26 |
| 4.6 | Safety Analyses (if not already covered as endpoint variables) | 26 |
| 4.6.1 | Exposure | 26 |
| 4.6.1.1 | Definitions and Derivations | 26 |
| 4.6.1.2 | Presentation | 26 |
| 4.6.2 | Adverse Events | |
| 4.6.2.1 | Definitions and Derivations | |
| 4.6.2.2 | Presentation | |
| 4.6.3 | Clinical Laboratory, Blood Sample | |
| 4.6.3.1 | Definitions and Derivations | 27 |

| STATISTICAL ANALYSIS PLAN | | AstraZeneca |
|---------------------------|---------------------------------|-------------|
| AZ-RU-00004 – ed. 3.0 | | 6-Aug-2024 |
| 4.6.3.2 | Presentations | 27 |
| 4.6.4 | Clinical Laboratory, Urinalysis | |
| 4.6.4.1 | Definitions and Derivations | |
| 4.6.4.2 | Presentations | |
| 4.6.5 | Other Laboratory Evaluations | 28 |
| 4.6.5.1 | Definitions and Derivations | |
| 4.6.5.2 | Presentations | 28 |
| 4.6.6 | Vital Signs | 28 |
| 4.6.6.1 | Definitions and Derivations | |
| 4.6.6.2 | Presentations | 28 |
| 4.6.7 | Electrocardiogram | |
| 4.6.7.1 | Definitions and Derivations | |
| 4.6.7.2 | Presentations | |
| 4.6.8 | Other Safety Assessments | 29 |
| 5 | INTERIM ANALYSIS | 29 |
| 6 | REFERENCES | 29 |
| 7 | APPENDIX | 29 |

# LIST OF ABBREVIATIONS

List abbreviations and definitions of specialized or unusual terms, measurements, or units. Examples are provided below. These can be modified at study level.

| Abbreviation or<br>Specialized Term | Definition |
|---|---|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| AR(1) | Autoregressive order 1 covariance matrix |
| AUC | Area Under Curve |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CS | Clinically Significant or Compound Symmetric covariance matrix |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| ECG | Electrocardiogram |
| ECT | Exercise Challenge Test |
| FAS | Full Analysis Set |
| FEV <sub>1</sub> | Forced Expiratory Volume in 1 second |
| FU | Follow Up |
| GAM | Generalized Additive Model |
| GCP | Good Clinical Practice |
| HR | Heart Rate |
| ICE | Intercurrent Event |
| ICH International Council for Harmonisation | |
| ICS | Inhaled Corticosteroid |
| IP | Investigational Product |
| IPD | Important Protocol Deviation |
| KM | Kaplan-Meier |
| LSMD | Least Squares Mean Difference |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model with Repeated Measures |
| NCS | Not Clinically Significant |
| PD | Protocol Deviation |
| PE | Physical Examination |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| SAE | Serious Adverse Event |

| Abbreviation or<br>Specialized Term | Definition |
|---|---|
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SOC | System Organ Class |
| TC | Telephone Call |
| TOEP | Toeplitz covariance matrix |
| UN | Unstructured covariance matrix |
| VS | Vital Signs |
| WHO Drug | World Health Organization Drug dictionary |

# **AMENDMENT HISTORY**

| CATEGORY Change refers to: | | Description of change | In line with CSP? | Rationale |
|---|---|---|---|---|
| N/A | 11/2/2023 | Initial approved SAP | N/A | N/A |
| Analysis sets 31/07/2024 e | | Name of enrolled/screened participants set is clarified Yes | | Clarification |
| Baseline characteristics | 31/07/2024 of smoking history is | | Yes | Clarification |
| 31/07/2024 | | Method of classification is added | Yes | Clarification after<br>meeting with<br>Study Clinical<br>Lead |
| Subgroup analysis 31/07/2 | | Wording is updated. GAM models are excluded | Yes | In order to be in line with the global study |
| Adverse events 31/07/2024 | | Some clarifications in analysis. | Yes | Clarification after<br>meeting with<br>Study Clinical<br>Lead |
| Other laboratory data 31/07/2024 | | Weight, height and<br>BMI will be presented<br>only in listings | Yes | Clarification after<br>meeting with<br>Study Clinical<br>Lead |
| Prior and concomitant medications Definitions and presentation of prior and concomitant medications medications was clarified | | Yes | Clarification after<br>meeting with<br>Lead Statistician | |
| Intercurrent event \ \ \ \ 06/08/2024 \ | | Intercurrent event strategy was clarified | Yes | Clarification after meeting with Lead Statistician |

# 1 INTRODUCTION

The purpose of the current statistical analysis plan (SAP) is a detailed description of basic principles of statistical analysis, description of methods used to analyse the primary and secondary endpoints, and other data obtained during the study.

This plan provides for compliance of the planned and conducted statistical analysis with the clinical study protocol (CSP), including the definition of datasets for analysis, transformations and calculations for endpoints, the required number of observations, etc. All discrepancies with the CSP should be clarified.

The current statistical analysis plan is prepared in compliance with:

- ICH harmonised tripartite guideline. Statistical principles for clinical trials (E9). Step 5 finalized guideline February 1998
- ICH harmonised tripartite guideline. Structure and Content of Clinical Study Reports (E3). Step 5 finalized guideline dated November 1995
- Good Clinical Practice of the Eurasian Economic Union, adapted by the decision of the Council of Eurasian Economic Commission on 3 November 2016, N 79
- Recommendation of the Board of the Eurasian Economic Commission No. 19 "On Guidelines for the Application of Biostatistics principles in Clinical trials of Medicinal Products", dated 3 November 2020

This SAP is based on version 1.0 of the CSP dated 29 August 2023. In case of future amendments to the protocol, the SAP may be modified to account for changes relevant to the statistical analysis.

# 2 CHANGES TO PROTOCOL PLANNED ANALYSES

This SAP is written in line with the current version of the CSP. All planned analyses correspond to the statistical section of the CSP.

## 3 DATA ANALYSIS CONSIDERATIONS

# 3.1 Timing of Analyses

It is planned to conduct only final analysis. It will be performed when all participants completed the study.

# 3.2 Analysis Populations

The following populations are defined:

Table 1. Populations for Analysis

| Population/analysis set | Description |
|---|---|
| Enrolled/screened participants set | All participants who sign the ICF. |
| Full analysis set (FAS) | All participants who are randomized to treatment and have at least one postdose, pre-exercise baseline and at least one corresponding post-dose postexercise FEV <sub>1</sub> measure at Visit 3 and/or Visit 4. |
| Safety analysis set | All participants who have received any amount of the study intervention. |

# 3.3 General Considerations

The data analyses will be conducted using SAS® System (SAS Institute Inc., Cary, NC), version 9.4 or higher.

In general, all data will be listed, sorted by treatment sequence (i.e. PT027/Placebo and Placebo/PT027) and participant, and when appropriate by visit number within participant.

Unless otherwise noted, data will be presented in tables by treatment sequence using descriptive statistics.

# **3.3.1** General Study Level Definitions

The below-mentioned general principles will be followed throughout the study:

- Descriptive statistics will be used for all variables, as appropriate.
  - Continuous variables will be summarised by the number of observations, mean, standard deviation, median, upper, and lower quartiles where indicated, minimum, and maximum by timepoint as appropriate.
  - Categorical variables will be summarised by frequency counts and percentages for each category. Unless otherwise stated, percentages will be calculated based on the analysis set population total by timepoint as appropriate.
- For continuous data, the mean, standard deviation and median are rounded to one additional decimal place compared to the original data. Minimum and maximum are displayed with the same accuracy as the original data.
- Time-to-event variables will be presented using the Kaplan-Meier (KM) methodology, including median time calculated from the KM curves.
- For categorical data, percentages are rounded to one decimal place with the exception of 100% which is presented as a whole number.

Only acceptable or usable spirometry values will be recorded in eCRF and included in the analyses and presented in tables, listings and figures. Values marked as usable will be utilized only in case if acceptable values are unavailable.

# 3.3.1.1 Period specific post-dose pre-exercise baseline

Post-dose pre-exercise baseline is defined as the FEV<sub>1</sub> result taken post-dose of randomized treatment and prior to the exercise challenge test conducted at Visit 3 and Visit 4 (approximately occurring 30 minutes post dose of IP, see CSP, Table 4).

The post-dose pre-exercise baseline is period specific and therefore will be calculated at each Visit 3 and Visit 4.

The post-dose pre-exercise baseline will be used to calculate the primary and secondary endpoints of changes from baseline.

# 3.3.1.2 Period specific pre-dose baseline

The period specific pre-dose baseline is defined as the spirometry measurement taken prior to dosing of randomized treatment, which should occur at 5 minutes pre-dose of IP (Table 4). The period specific pre-dose baseline will be calculated separately at Visit 3 and Visit 4.

The period specific pre-dose baseline will be included as a covariate in parametric analyses of the primary and secondary endpoints.

The period specific pre-dose baseline will additionally be used to calculate changes from baseline in safety endpoints of vital sign parameters and ECG parameters.

# 3.3.1.3 Average pre-dose baseline

The average pre-dose baseline will be calculated as the average of the non-missing period specific pre-dose baseline result for each subject. The average pre-dose baseline will be included as a covariate in parametric analyses of the primary and secondary endpoints.

# 3.3.1.4 Absolute and percent change from baseline

Absolute change from baseline outcome variables is computed as:

Absolute change from baseline =  $(post-baseline\ value-baseline\ value)$ .

Percent change from baseline is computed as:

Percentage change from baseline =  $[(post-baseline \ value - baseline \ value) / baseline \ value] * 100%.$ 

If either the post-baseline value or the baseline value is missing, then the absolute/percent change from baseline value will also be set to missing.

#### 3.3.1.5 Percentage fall from post-dose pre-exercise baseline FEV<sub>1</sub>

Percentage fall from post-dose pre-exercise baseline  $FEV_1$  will be used to calculate primary and secondary lung function endpoints and is defined as:

Percentage fall from post-dose pre-exercise baseline = [(post-dose pre-exercise baseline value - post-exercise value) / post-dose pre-exercise baseline value]  $\times$  100%.

The percentage fall from post-dose pre-exercise FEV<sub>1</sub> will be calculated at each postexercise timepoint at Visits 2, 3 and 4.

If either the post-baseline value or the baseline value is missing, then the percentage fall from baseline value will also be set to missing.

#### 3.3.1.6 Crossover difference in maximum percentage fall of FEV<sub>1</sub>

Crossover difference in maximum percentage fall of FEV<sub>1</sub> will be calculated for each participant as difference of maximum percentage fall of FEV<sub>1</sub> registered in period of PT027 administration and maximum percentage fall of FEV<sub>1</sub> registered in period of Placebo administration.

#### 3.3.2 Visit Window

Due to the design of this trial, there will be no visit windowing applied other than the identification of baseline.

#### 3.3.3 **Handling of Unscheduled Visits**

Retest and reassessment of spirometry will be registered as unscheduled visits. If some retests will be registered after Visit 3 and before Visit 4 then the latest result will be included in the analysis as result of Visit 3. If some retests will be registered after Visit 4 then the latest result will be included in the analysis as result of Visit 4. All other results will be presented only in listings. Other unscheduled and early discontinuation measurements will not be included in by-visit summaries.

#### 3.3.4 **Multiplicity/Multiple Comparisons**

For purposes to demonstrate statistically significant superiority of the IMP, the following comparison sequence will be conducted:

- Primary endpoint: the maximum percentage fall from post-dose, pre-exercise baseline in forced expiratory volume in 1 second (FEV<sub>1</sub>) observed up to 60 minutes post-exercise challenge
- 2. Secondary endpoint: the percentages of subjects with a maximum percentage fall in FEV<sub>1</sub> post-exercise challenge of <10%

If 1<sup>st</sup> comparison is significant ie obtained 2-sided p-value < 0.05, then 2<sup>nd</sup> comparison will be reported as significant if corresponding obtained 2-sided p-value < 0.05.

#### 3.3.5 **Handling of Protocol Deviations in Study Analysis**

Protocol deviations will be collected, reviewed, and reconciled throughout the study. Important protocol deviations (IPDs) will be identified from the complete set of protocol deviations. IPDs are those which may significantly impact the completeness,

accuracy, or reliability of the study data or that may significantly affect a participant's rights, safety, or wellbeing.

All decisions on importance will be made throughout the study and finalised before clinical data base lock.

#### 3.3.6 **Missing Data**

Safety assessments of the form of "<x" (ie, below the lower limit of quantification) or ">x" (ie, above the upper limit of quantification) are imputed as "x" in the calculation of summary statistics but are displayed as "<x" or ">x" in the listings.

For missing start dates for adverse events (AEs) and medications/procedures, the following rules are applied:

- Missing day: Impute the first of the month unless the month is the same as month of the first dose of study drug and the end date is on or after the first dose of study drug or ongoing then impute first dose date
- Missing day and month: Impute 01 January unless year is the same as first dose date and the end date is on or after the first dose of study drug or ongoing then impute first dose date.
- Completely missing date:
  - o For AEs and treatment identified as prior to study start in the eCRF (i.e. end date before day of first dose): Impute the day before first dose date unless the end date is prior to this in which case impute the date the patient was enrolled.
  - o For treatment not identified as prior to study start in the eCRF, no imputation will be performed. For an AE not identified as prior to study start, the date of first dose will be imputed.

An imputed start date of an AE must be prior to the end date of the AE.

For missing stop dates of AEs or medications/procedures, the following rules are applied:

- Missing day: Impute the last day of the month unless month is the same as month of study discontinuation, then impute as study discontinuation date. For prior medications impute date of informed consent if month is the same as month informed consent was provided.
- Missing day and month: Impute 31 December unless year is the same as year of study discontinuation then impute study discontinuation date. For prior medications impute date of informed consent if year is the same as month informed consent was provided.

- Completely missing: If an AE/medication has a completely missing end date then it is treated as ongoing unless the outcome is stated in the eCRF as recovered/resolved for AEs or treatment continues stated as "No" for medications.
  - o If the AE/medication is not ongoing (as identified in the eCRF), then the stop date will be imputed by the date of study discontinuation.
  - o For stopped medication, if the medication is marked as prior and start date is prior to first dose date, then impute the date of the day before first dose.
  - If the medication started on or after first dose date, then impute the date of study discontinuation.

The imputation of dates for AEs and medications are used to determine if an AE is treatment emergent and whether a medication is concomitant. Flags are retained in the database indicating where any programmatic imputation has been applied, and in such cases, any durations are not calculated.

For time to event endpoints, dropouts and missing data are handled according to the censoring rules detailed within the relevant sections for the endpoint.

Other rules for handling missing data are described under the derivation rules for that particular variable.

#### STATISTICAL ANALYSIS 4

This section provides information on definitions, derivation and analysis/data presentation per domain.

#### 4.1 **Study Population**

The domain study population covers subject disposition, analysis sets, protocol deviations, demographics, baseline characteristics medical history, prior and concomitant medication and study drug compliance.

#### 4.1.1 **Subject Disposition and Completion Status**

#### 4.1.1.1 **Definitions and Derivations**

Participants disposition and completion status will be comprised of the following:

- Enrolled participants;
- Non-randomized participants (screen failures);
- Randomized participants;
- Participants who were randomized but no dosed with reasons;
- Participants who were randomized and treated on 1<sup>st</sup> period;
- Participants who were randomized and treated on 2<sup>nd</sup> period;

- Participants who were randomized and treated with PT027
- Participants who were randomized and treated with placebo
- Randomized participants who completed FU visit.
- Randomized participants who withdrew from the study with reasons

## 4.1.1.2 Presentation

Number and percentage of participants in each category will be reported by treatment sequence for Enrolled/Screened Participants Set.

# 4.1.2 Analysis Sets

# **4.1.2.1 Definitions and Derivations**

Refer to Section 3.2 for definition of analysis sets:

- Enrolled/Screened Participants Set
- Full Analysis Set
- Safety Analysis Set

#### 4.1.2.2 Presentation

The number of participants included in each analysis set will be reported by treatment sequence for Enrolled/Screened Participants Set. In addition, for each analysis set, the number of participants excluded, including the reasons, will be reported, if applicable.

## 4.1.3 Protocol Deviations

## **4.1.3.1 Definitions and Derivations**

A detailed list of possible important protocol deviations (IPDs) and the process for reviewing them by the clinical study team will be outlined in the Protocol Deviation plan (PD plan).

The medical and statistical team members will review the protocol deviation categories in a blinded fashion before the clinical database lock and be classified as important per the PD plan.

At a minimum, the following deviations categories will be included for review and classified as important for the evaluation and implementation of the study:

- Inclusion Criteria Deviations
- Exclusion Criteria Deviations
- Discontinuation Criteria for study product met but participant not withdrawn from study treatment
- Discontinuation Criteria for overall study withdrawal met but participant not withdrawn from study
- Investigational Product Deviation
- Excluded Medications taken

- Deviations to study procedure
- Other Important Protocol Deviations

## 4.1.3.2 Presentation

The number and percentage of participants with IPDs will be provided per protocol deviation category. The summary will be based on the Safety Analysis Set.

All important protocol deviations will be presented in a listing.

# 4.1.4 Demographics

#### 4.1.4.1 Presentation

Following demographic characteristics will be summarized for all participants in the Safety Analysis Set:

- Age
- Age group
  - o <65 years
  - o ≥65 years
- Sex
- Race
- Ethnic group

# 4.1.5 Baseline Characteristics

# 4.1.5.1 Presentation

Following baseline characteristics will be summarized for all participants in the Safety Analysis Set:

- Weight (kg)
- Height (cm)
- Body mass index (BMI, kg/m<sup>2</sup>)
- Maximal HR results during Exercise Test for visits 1 and 2
- Smoking history
- Results of spirometry on Visits 1 and 2
- Results of spirometry on Visit 3 prior randomization

# 4.1.6 Disease Characteristics

Disease characteristics will be presented for the Safety Analysis Set.

# 4.1.6.1 Definitions and Derivations

The following characteristics will be collected:

- Allergen asthma trigger
- Aspirin asthma trigger
- Exercise asthma trigger
- Other asthma trigger

The time since diagnosis of asthma (years) will be calculated as:

(Date of first dose of randomized treatment (Visit 3) - Date of diagnosis of asthma)/365.25.

Partial dates for the above calculations will be handled as per Section 3.3.6.

#### 4.1.6.2 Presentation

Disease characteristics will be presented in a table with descriptive statistics and in a listing.

# 4.1.7 Medical History and Concomitant Disease

## 4.1.7.1 Definitions and Derivations

Medical history and relevant surgical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 26.1 or later. The version used will be indicated in the tables and listings.

Any medical history which is ongoing at time of informed consent will be considered as current medical history, otherwise it is considered as past medical history.

Clinically significant abnormal physical examination findings at screening will be recorded as adverse events

## 4.1.7.2 Presentation

Past and current medical history will be grouped by MedDRA System Organ Class (SOC) and Preferred Term (PT) and summarized in the Safety Analysis Set as number and percentage of participants in each treatment sequence.

Also past and current medical history will be presented in listings.

#### 4.1.8 Prior and Concomitant Medications

# 4.1.8.1 Definitions and Derivations

**Prior medication:** all prescripted drugs, herbal products, vitamins, minerals, and over-the-counter medications with end date within 3 months before date of randomization.

**Concomitant medications:** all medications with start date on or after date of randomization, or with end date after date of randomization or ongoing at the time of the follow-up telephone call (TC).

If a medication has start date before date of randomization and end date after date of randomization or ongoing the follow-up telephone call (TC), so this medication will be considered as prior and as concomitant, therefore it will be presented in both corresponding tables.

#### **Restricted Medications**

As described in Table 8 of the CSP.

#### **Prohibited Medications**

As described in Table 8 of the CSP. Medications will be classified as prohibited or not on the medical review.

# **Rescue Medications**

AstraZeneca will supply rescue medication – Ventolin® (salbutamol, SABA), 100 µg metered dose inhaler, to the study site.

For the purpose of inclusion in prior or concomitant mediation, incomplete medication start and stop dates will be imputed as detailed in Section 3.3.6.

#### 4.1.8.2 **Presentation**

All medications will coded using World Health Organization Drug dictionary (WHO Drug) version Sep 2023 B3 or later. The version used will be indicated in the data summaries and listings. Medications will be presented in the Safety Analysis Set.

Prior and concomitant medications will be presented in separate outputs.

The number and percentage of participants receiving prior or concomitant medication (by ATC classification system codes and generic name) will be presented by treatment sequence.

Additionally, prior and concomitant medications will be listed. The listing of concomitant medications will include reason for use, start and end dates of administration, dosage information including dose, frequency and route.

Restricted medications also will be listed. The listing will include date and time of SABA administration and date and time of consequent planned FEV<sub>1</sub> testing procedures.

Events of prohibited medication administration will be registered and presented as protocol deviations (Section 4.1.3).

Data on rescue medication administrations will be listed. The listing will include date, time of administration, name and dosage regimen.

#### 4.1.9 **Study Drug Compliance**

Not applicable for this study.

#### 4.2 **Endpoint Analyses**

This section covers details related to the endpoint analyses such as primary, secondary, other endpoints including sensitivity and supportive analyses.

Descriptive statistics and analysis results (if applicable) will be presented by treatment, unless otherwise specified.

Examples of SAS code implemented efficacy analysis models presented in corresponding sections. These codes can be updated, for example, in order to obtain necessary statistics of a model.

| Statistical category | Endpoint | Analysis<br>Set | Intercurrent event strategy | Population<br>level summary<br>(analysis) | Details<br>in<br>section |
|---|---|---|---|---|---|
| with placeb | | | (budesonide/albuterol) metered<br>e dose on exercise-induced brond | | |
| Primary | The maximum percentage fall from post-dose, pre-exercise baseline in forced expiratory volume in 1 second (FEV <sub>1</sub> ) observed up to 60 minutes post-exercise challenge | Full<br>Analysis<br>Set | Intercurrent event defined as rescue medication administration prior to the first spirometry reading. Only FEV <sub>1</sub> results prior to rescue therapy (within the study visit) will be included in the analyses. A while on treatment strategy will be used such that missing values will be assumed missing at random (MAR) and handled by the direct likelihood methods of the mixed effects model. Missing data not preceded by an intercurrent event, such as subjects who withdraw from study will be assumed to be MAR. | Difference of means between treatments | 4.2.1 |
| compared w | | | of PT027 (budesonide/albutero)<br>ter a single dose on exercise-ind | | |
| Secondary | The percentages of subjects with a maximum percentage fall in FEV <sub>1</sub> post-exercise challenge of <10% and <20%, respectively | Full<br>Analysis<br>Set | While on treatment strategy will be applied as a primary strategy: only FEV <sub>1</sub> results prior to administration of rescue medication (within | The percentage fall will be calculated relative to the pre-exercise FEV <sub>1</sub> assessment at | 4.2.2 |

| Statistical | | Analysis | | Population<br>level summary | Details<br>in |
|---|---|---|---|---|---|
| category | Endpoint | Set | Intercurrent event strategy | (analysis) | section |
| | | | the study visit) will be analysed. Composite strategy will be used for purposes of a supplementary analysis: articipants who used rescue medication administration prior to the first spirometry reading will be analysed as non-responders | the respective visit. The measure of interest is the odds ratio between PT027 and Placebo for each threshold separately (<10% and <20%). | |
| Secondary | The percentage fall from post-dose, pre-exercise baseline in FEV <sub>1</sub> at each timepoint within 60 minutes post-exercise challenge | Full<br>Analysis<br>Set | Hypothetical strategy will be used for analysis of this endpoint: only FEV <sub>1</sub> results prior to administration of rescue medication (within the study visit) will be included in the analyses, missing values will be utilized in the analysis by using the mixed model with repeated measures (MMRM). | The measure of interest is the percentage fall from baseline in FEV <sub>1</sub> at each timepoint within 60 minutes post-exercise challenge. | 4.2.3 |
| Secondary | Post-exercise FEV1<br>area under the curve<br>from 0 to 30 minutes<br>(AUC <sub>0-30min</sub> ) | Full<br>Analysis<br>Set | While on treatment strategy will be applied: only the FEV <sub>1</sub> AUC <sub>0-30min</sub> measurements prior to administration of rescue medication will be included in the analyses. | The measure of interest is the difference between treatments in the post-exercise FEV <sub>1</sub> AUC <sub>0</sub> . | 4.2.4 |
| Secondary | Time to recovery, defined as the time from completionof the exercise challenge to the first measured post-exercise challenge FEV <sub>1</sub> value within 10% of the post-dose, pre-exercise challenge baseline FEV <sub>1</sub> | Full<br>Analysis<br>Set | While on treatment strategy will be applied: only FEV <sub>1</sub> results prior to administration of rescue medication (within the study visit) will be included in the analyses | The measure of interest is the median of the time to recovery. | 4.2.5 |
| <b>Objective 3:</b> To assess the safety and tolerability of PT027 (budesonide/albuterol) metered-dose inhaler as compared with placebo metered-dose inhaler after a single dose in adult participants with asthma. | | | | | |
| | Safety and | | | The measure of | |
| Safety | tolerability will be evaluated in terms of: • AEs • SAEs • AEs lead to discontinuation. | Safety<br>Analysis<br>Set | All data will be analysed | interest is<br>frequencies and<br>percentages of<br>participants with<br>reported AEs | 4.6.2 |

| Set | Intercurrent event strategy | (analysis) | section |
|----------------------|-----------------------------|------------|------------|
| CGs will ed in terms | | | |
| | d in terms | d in terms | d in terms |

# 4.2.1 Primary Endpoint

# 4.2.1.1 Definition

The primary variable is the maximum percentage fall of FEV<sub>1</sub> available in the post-exercise 60-minute assessment period prior to the use of rescue medication, from FEV<sub>1</sub> value measured after study treatment and prior to the exercise. It will be calculated at Visit 3 and Visit 4.

#### 4.2.1.2 Derivations

The fall from post-dose, pre-exercise baseline in FEV<sub>1</sub> will be calculated at each post-exercise FEV<sub>1</sub> assessment time point within Visits 3 and 4 as described in Section 3.3.1.

The post-dose, pre-exercise baseline FEV<sub>1</sub> assessment is expected to occur 30 minutes after administration of IP and 5 minutes prior to the exercise challenge within Visits 3 and 4.

The percentage fall in FEV<sub>1</sub> will be calculated as difference from to the post-exercise value to the pre-exercise value at each measurement during the 60-minute assessment period divided by the pre-exercise value and presented in percents within Visits 3 and 4.

The maximum percentage fall available in the 60-minute assessment period, prior to the use of rescue medication, will be calculated at Visit 3 and Visit 4.

# 4.2.1.3 Handling of Dropouts and Missing Data

Values of FEV<sub>1</sub> obtained after rescue medication and missing values will not be imputed.

# 4.2.1.4 Primary Analysis of Primary Endpoint

The primary analysis will be performed in the FAS. Only data prior to the occurrence of an intercurrent event (ICE) will be included in the analysis in accordance with the WoT strategy.

The primary efficacy endpoint will be analyzed with a mixed effect model including categorical fixed effects for treatment, treatment period and treatment sequence. Continuous covariates include period-specific pre-dose baseline  $FEV_1$  and average pre-dose baseline  $FEV_1$  (as defined in Section 3.3.1.3) in order to eliminate cross-level bias whilst using pre-treatment baselines. Also, a random subject within treatment sequence effect will be specified.

Post-dose, pre-exercise baseline FEV<sub>1</sub> will be defined as the 30-minute post-dose value, i.e., 5 minutes before exercise challenge, at each visit for the respective treatment. The period-specific pre-dose baseline FEV<sub>1</sub> will be calculated separately at Visit 3 and Visit 4 as the pre-dose result, approximately 5 minutes prior to dosing. The average pre-dose baseline FEV<sub>1</sub> will be calculated as the mean of the period-specific pre-dose FEV<sub>1</sub> baselines. Estimated treatment differences and 95% confidence intervals (CIs) will be provided.

Applied significance level (alpha): 0.05 (using a 2-sided test).

Additionally, least squares mean estimates, 95% confidence intervals and associated p-values of the treatment difference will be calculated for the subgroups of clinical interest by additionally adjusting for background therapy (ICS or no ICS) and background therapy\*treatment group interaction in the mixed model.

A forest plot will be created showing the difference in least squares mean estimates and associated 95% confidence intervals for the Overall, ICS and non-ICS subgroups.

Model results as well as descriptive statistics will be presented in tables. Figure for adjusted means and 95% CIs will be presented.

All data will be listed.

# 4.2.1.5 Sensitivity Analyses of the Primary Endpoint

Missing results for maximum percentage fall in  $FEV_1$  are unlikely (i.e., rescue medication prior to the collection of the 5 minutes measure) and will be assumed to be missing at random. Sensitivity analysis will be conducted to explore the robustness of the primary analysis with respect to this missing data assumption. This analysis will be conducted in supportive purposes.

Data that are missing will be imputed using reference-based imputation. Participants with a missing maximum percentage fall in the 60-minute assessment period, for any visit, will be imputed using the least squares mean estimate of the maximum percentage fall in the Placebo treatment from a mixed model as specified in Section 4.2.1.4, using the observed data. After imputation the dataset of complete data, will be analyzed using the same model as descripted in Section 4.2.1.4.

Model results as well as descriptive statistics will be presented in tables. Figure for adjusted means and 95% CIs will be presented.

All data will be listed.

# 4.2.2 Secondary Endpoint: the percentages of subjects with a maximum percentage fall in FEV<sub>1</sub> of <10% and <20%

#### 4.2.2.1 Definition

Protection against EIB will be defined having a maximum percentage fall in FEV<sub>1</sub> post-exercise change under the corresponding threshold values (<10% and <20%)

## 4.2.2.2 Derivations

Derivation will be completely based on comparing primary efficacy variable (described in Section 4.2.1.1) and threshold values of 10% and 20%.

For each threshold value a participant will be considered as protected patient (responder) if their maximum percentage fall in FEV<sub>1</sub> post-exercise change was less than the threshold value. Therefore two different types of responders will be analysed.

# 4.2.2.3 Handling of Dropouts and Missing Data

Participants with missing maximum percentage fall will not be included in the primary analysis.

# 4.2.2.4 Primary Analysis of Secondary Endpoint

The odds of being protected against EIB will be analyzed using a generalized linear mixed model with logit link function to compare the treatments. Two separate models will be presented for each two types of responders (participants protected against EIB) as described in Section 4.2.2.2.

The models will be adjusted with fixed effects for treatment, treatment period and treatment sequence, period specific pre-dose baseline  $FEV_1$  and average pre-dose baseline  $FEV_1$  as continuous covariates, and a random subject within treatment sequence effect. The odds ratio and 95% CI will be reported for pairwise treatment comparisons.

Model results as well as descriptive statistics will be presented in tables and figures. All data will be listed.

# 4.2.2.5 Supplementary Analysis of Secondary Endpoint

The suplementary analysis of this endpoint will be performed using the same models as in the primary analysis but participants who didn't withdraw the study prematurely and had missing maximum percentage fall will be analysed as non-responders.

Model results as well as descriptive statistics will be presented in tables and figures. All data will be listed.

# 4.2.3 Secondary Endpoint: the percentage fall in FEV<sub>1</sub> from post-dose, pre-exercise at each timepoint within 60 minutes post-exercise

# 4.2.3.1 Derivations

Described in Section 4.2.1.2.

# 4.2.3.2 Handling of Dropouts and Missing Data

Described in Section 4.2.1.2.

# 4.2.3.3 Primary Analysis of Secondary Endpoint

An analysis of percentage fall in  $FEV_1$  post-exercise challenge will be conducted using methods as per the primary analysis, with an additional adjustment for planned time point in the repeated measures model. The covariance within subject-periods will be Unstructured (UN) over the time points. In case of impossible to build the model due to divergence, the following variants of the covariance matrix will be sequentially tested: Compound Symmetric (CS), Autoregressive, order 1 (AR(1)), Toeplitz (TOEP).

Only  $FEV_1$  results prior to administration of rescue therapy (within the study visit) will be included in the analyses.

Model results as well as descriptive statistics will be presented in tables. Figures for adjusted means and 95% CIs as well as unadjusted means and 95% CIs will be presented.

All data will be listed.

# 4.2.4 Secondary Endpoint: post-exercise FEV<sub>1</sub> area under the curve from 0 to 30 minutes

## 4.2.4.1 Definition

Post-exercise  $FEV_1$  area under the curve (AUC) from 0 to 30 minutes will be defined on the base of changes from baseline in  $FEV_1$  as defined in Section 4.2.1.2 for time points planned up to 30 minutes after the test.

#### 4.2.4.2 Derivations

Post-exercise FEV<sub>1</sub> area under the curve from 0 to 30 minutes (FEV<sub>1</sub> AUC<sub>0-30min</sub>) will be derived for the changes from the post-dose, pre-exercise baseline using the trapezoidal rule and will be normalized by dividing by the actual time (in minutes) from the exercise challenge test to the last included measurement, scheduled at 30 minutes post-exercise challenge at each of Visits 3 and 4. Only FEV<sub>1</sub> results prior to the use of rescue medication will be considered when calculating FEV<sub>1</sub> AUC<sub>0-30min</sub>.

$$AUC_{0-30 \ minutes} = \frac{1}{t_N - t_0} \times \sum_{i=1}^{N} \frac{(y_{i-1} + y_i) \times (t_i - t_{i-1})}{2}$$

For FEV<sub>1</sub> change from baseline results  $y_i$  recorded  $t_i$  minutes after the exercise challenge test (actual clock time) at i=0,1,2,...,N actual timepoints. If all post-exercise timepoints are available, then N=4,  $t_0$  corresponds to the end time of the exercise challenge test and  $y_0=0$ . Only FEV<sub>1</sub> results of 'acceptable' or 'borderline acceptable' (investigator assigned) quality will be used in the derivation of FEV<sub>1</sub> AUC<sub>0-30min</sub>. If a FEV<sub>1</sub> result is missing or recorded in the database, but assigned an

'unacceptable' quality grade at the scheduled assessment, then the assessment will be excluded from the calculation of  $FEV_1$   $AUC_{0-30min}$ . To calculate  $FEV_1$   $AUC_{0-30\,min}$ , there must be at least 1 non-missing post-dose  $FEV_1$  within 0 to 30 minutes post-dose. Missing  $FEV_1$  post-dose measures will not be imputed.

# 4.2.4.3 Handling of Dropouts and Missing Data

Values of FEV<sub>1</sub> obtained after rescue medication and missing values will not be imputed. Missing actual times for non-missing change from baseline values will be replaced with planned times.

# 4.2.4.4 Primary Analysis of Secondary Endpoint

The endpoint will be analyzed using the same approach as described in Section 4.2.1.4.

# 4.2.5 Secondary Endpoint: time to recovery

## 4.2.5.1 Definition

Recovery will be defined as return of post-exercise changes of the FEV<sub>1</sub> within 10% interval of the value recorded at the post-dose, pre-exercise baseline.

#### 4.2.5.2 Derivations

Time to recovery at each of Visits 3 and 4 will be derived as the time (in minutes) post-exercise challenge in which the FEV<sub>1</sub> result returns to within 10% of the value recorded at the post-dose, pre-exercise baseline.

The post-dose, pre-exercise baseline  $FEV_1$  assessment and percentage fall in  $FEV_1$  will be calculated as described in Section 4.2.1.2, at Visit 3 and Visit 4 separately.

# 4.2.5.3 Handling of Dropouts and Missing Data

Missing values of FEV<sub>1</sub> and times of measurements will not be imputed.

# 4.2.5.4 Primary Analysis of Secondary Endpoint

The median time to recovery will be reported descriptively by treatment. P-values will be calculated using a Prescott's period-adjusted sign test, based on categorizing subjects into period preferences (Senn S 1993).

# Censoring rules:

- If a participant has not observed a fall greater than 10% of the post-dose preexercise baseline in their post-exercise challenge test by 60 minutes, they will be left censored at 0 minutes.
- Participants who have any rescue medication administered during the post-dose assessments will be censored at the time of receiving rescue medication.
- Participants who do not recover to within 10% of the post-dose, pre-exercise baseline will be censored at their last assessment.

# 4.2.6 Other Endpoints

Not applicable.

# 4.2.7 Subgroup Analyses

The assessment of treatment effect will also be investigated for primary endpoint (described in Section 4.2.1) and first secondary endpoint (described in Section 4.2.2) in the other clinically important subgroups described in Table:

Table 3. Subgroup Analyses

| Group | Subgroup |
|-----------------------------|-------------------------------------|
| Sex | Male |
| | Female |
| Age group (years) | Adults: ≥ 18 - < 65 |
| | Elderly: >= 65 |
| BMI (kg/m2) | Median value cut-off <sup>[1]</sup> |
| Baseline FEV <sub>1</sub> % | Median value cut-off <sup>[1]</sup> |

[1] Subgroup will be categorized into 2 groups defined by the median value observed at baseline. Baseline FEV1 % for grouping purposes here will be pre-dose baseline FEV1 % predicted normal at Visit 3.

For all subgroup analyses, if there are less than 10 subjects/events available within a subgroup and at least 5 subjects with data available per treatment group under comparison, or the model does not converge, then only descriptive (summary) statistics will be presented. Subgroup analyses will be further broken down into the overall population, and ICS and non-ICS populations. Subjects with insufficient data to be allocated to a subgroup category will be excluded from the subgroup analyses.

Model results as well as descriptive statistics will be presented in tables. Figures for adjusted means and 95% CIs will be presented.

Forest plots will be produced showing the least squares mean difference and associated 95% confidence intervals within each subgroup for the primary endpoint of maximum percentage fall from post-dose, pre-exercise baseline in FEV<sub>1</sub>.

All data will be listed.

# 4.3 Pharmacodynamic Endpoint(s)

Not applicable

# 4.4 Pharmacokinetics

Not applicable

# 4.5 Immunogenicity

Not applicable

# **4.6** Safety Analyses (if not already covered as endpoint variables)

The domain safety covers exposure, adverse events, clinical laboratory, vital signs, and ECG.

Tables and listings will be provided for the Safety Analysis Set.

# 4.6.1 Exposure

# **4.6.1.1 Definitions and Derivations**

Participants will have single administration of placebo at the screening period and single administrations of placebo or PT027 (depending of randomization) on each of both study periods.

#### 4.6.1.2 Presentation

Number and percentage of participants who received both treatments and who didn't receive the second treatment (Visit 4) with reasons will be presented by treatment sequence. Placebo administration on Visit 2 will not be accounted.

All data on exposure will be listed.

## 4.6.2 Adverse Events

## 4.6.2.1 Definitions and Derivations

AEs will be coded by System Organ Class (SOC) and Preferred Term (PT) using the latest version of the MedDRA dictionary.

#### 4.6.2.2 Presentation

AEs started before time of study treatment on Visit 3 will be considered as pretreatment AEs and will be presented in a separate listing.

AEs of participants from A/B treatment sequence registered in period from time of study treatment on Visit 3 to time of study treatment on Visit 4 and AEs of participants from B/A treatment sequence registered after time of study treatment on Visit 4 will be considered as AEs of PT027. If participant from A/B treatment sequence didn't receive study treatment on Visit 4, then all AEs occurred after time of study treatment on Visit 3 will be considered as AEs of PT027.

AEs of participants from B/A treatment sequence registered in period from time of study treatment on Visit 3 to time of study treatment on Visit 4 and AEs of participants from A/B treatment sequence registered after time of study treatment on Visit 4 will be considered as AEs of Placebo. If participant from B/A treatment sequence didn't receive study treatment on Visit 4, then all AEs occurred after time of study treatment on Visit 3 will be considered as AEs of placebo.

The following tables by IP will be presented:

- Overall table for AEs
- AEs by SOC and PT
- SAEs by SOC and PT
- AEs related to study intervention by SOC and PT
- SAEs related to study intervention by SOC and PT
- AEs by SOC and PT, by severity
- AEs by SOC and PT, by outcome
- SAEs by SOC and PT, by outcome
- AEs by SOC and PT, by action taken with IMP
- SAEs by SOC and PT, by action taken with IMP
- AEs leading to discontinuation of study intervention, by SOC and PT
- AEs by SOC and PT caused participant to withdraw from the study

The following lisitngs will be provided:

- Pre-treatment AEs
- AEs (excluding the pre-treatment AEs)
- SAEs (excluding the pre-treatment AEs)
- AEs with fatal outcome

# 4.6.3 Clinical Laboratory, Blood Sample

# **4.6.3.1 Definitions and Derivations**

Blood samples for determination of clinical chemistry and hematology will be taken only at Screening (Visit 1). Additional safety samples may be collected if clinically indicated at the discretion of the investigator. Detailed list of parameters is presented in the CSP, Section 8.2.5.

#### 4.6.3.2 Presentations

Measured values at Screening will be presented with descriptive statistics as planned in Section 3.3.1 by treatment sequence in tables.

All data on blood samples will be presented in listings.

# 4.6.4 Clinical Laboratory, Urinalysis

# 4.6.4.1 Definitions and Derivations

Urine samples for urinalysis will be taken only at Screening (Visit 1). Detailed list of parameters is presented in the CSP, Section 8.2.5.

## 4.6.4.2 Presentations

Results of urinalysis will be presented in a listing.

# 4.6.5 Other Laboratory Evaluations

# 4.6.5.1 Definitions and Derivations

A serum pregnancy test ( $\beta$ -human chorionic gonadotropin [ $\beta$ -hCG]) will be performed at Visit1, 4 and PDV; urine  $\beta$ -hCG test will be performed at Visit 3 (for women of childbearing potential only).

Urine samples will be taken during Visits 1-4 for drugs of abuse and cotinine testing. The analysis will be carried out using test strips. The list of psychoactive agents for testing includes marijuana, benzodiazepines, barbiturates, opiates, methadone, phencyclidine, cocaine, amphetamines.

Also, during Visits 1-4 alcohol detection test will be performed using breathalyser.

#### 4.6.5.2 Presentations

All data of these additional laboratory tests will be presented in listings.

# 4.6.6 Vital Signs

#### 4.6.6.1 Definitions and Derivations

Vital sings will be collected according to the Schedule of Activities: CSP, Section 1.3.

#### 4.6.6.2 Presentations

SBP, DBP and HR will be presented with descriptive statistics in tables using the following approach:

For Visit 1: measured values and changes for values on 20, 40 and 60 minutes after the test from values on 50 minutes before the test. Grouping by treatment sequence.

For Visit 2: measured values and changes for values on 20, 40 and 60 minutes after the dosing from values on 50 minutes before the dosing. Grouping by treatment sequence.

For visits 3 and 4: measured values and changes for values on 20, 40 and 60 minutes after the dosing from values on 50 minutes before the dosing. Grouping by treatment.

For visits 3 and 4: maximal HR during ECT. Grouping by treatment.

Treatments will be summarized using the same algorithm as described for AEs in Section 4.6.2.2.

Also all data on vital signs, including weight, height and BMI, will be presented in a listing.

# 4.6.7 Electrocardiogram

# **4.6.7.1 Definitions and Derivations**

Electrocardiogram will be performed according to the Schedule of Activities: CSP, Section 1.3.

#### 4.6.7.2 Presentations

Continuous parameters of ECG will be presented using the following approach:

For each visit: measured values and changes for values on 45 minutes after the test from values on 50 minutes before the test.

Interpretation of ECG as nominal parameter will be presented in shift tables for values on 50 minutes before the test and for values on 45 minutes after the test. Number and percentages of participants with values: Normal, Borderline, Abnormal NCS and Abnormal CS will be presented.

For visits 1 and 2, for continuous parameters and interpretation grouping will be performed by treatment sequence.

For visits 3 and 4, for continuous parameters and interpretation grouping will be performed by treatment. Treatments will be summarized using the same algorithm as described for AEs in Section 4.6.2.2.

Also all data on vital signs will be presented in a listing.

# 4.6.8 Other Safety Assessments

Not Applicable

# 5 INTERIM ANALYSIS

Not Applicable

## 6 REFERENCES

- ICH harmonised tripartite guideline. Statistical principles for clinical trials (E9). Step 5 finalized guideline February 1998;
- ICH harmonised tripartite guideline. Structure and Content of Clinical Study Reports (E3). Step 5 finalized guideline dated November 1995;
- Good Clinical Practice of the Eurasian Economic Union, adapted by the decision of the Council of Eurasian Economic Commission on 3 November 2016, N 79.
- Senn S, Cross-over Trials in Clinical Research. Wiley, Chichester.1993.

# 7 APPENDIX

Not Applicable

# Signature Page for CC System v1.0 BREATH\_SAP\_3.0

| Approve: Document Level Task | val |
|------------------------------|-------------------------------|
| Verdict: Approved | 06-Aug-2024 08:06:20 GMT+0000 |
| Approve: Document Level Task | Approval |
| Verdict: Approved | 06-Aug-2024 08:12:54 GMT+0000 |

Signature Page for CC System v1.0 BREATH\_SAP\_3.0